CLINICAL TRIAL: NCT07038928
Title: A Multicentre Observational Study on Treatment Approaches and HER2 Positive Status Prevalence in Different Stages of Bladder Cancer and PD-L1-positive Status in Metastatic Bladder Cancer in Russian Federation
Brief Title: TReatment Approaches and bIomarkers preValence in bladdEr Cancer in RuSsian Federation
Acronym: RIVERS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00057
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Patients with NMIBC: Non-muscle-invasive bladder cancer
- Patients with MIBC: Muscle-invasive bladder cancer
- Patients with mBC: Metastatic bladder cancer

SUMMARY:
A multicentre observational study on treatment approaches and HER2 positive status prevalence in different stages of bladder cancer and PD-L1-positive status in metastatic bladder cancer in Russian Federation

DETAILED DESCRIPTION:
This is an observational study entailing primary and secondary data collection. As an observational, this study does not imply any intervention into a routine clinical practice, including choice of treatment modality or additional diagnostic methods. Epidemiologic methods and descriptive analysis will be used for data collection and evaluation of all endpoints and measurements of interest.

It will be a multicentre study. Planned number of study sites is about 30 oncological centres performing specialised treatment and follow-up of patients with urothelial bladder cancer in different regions of Russia. Planned study population consists of approximately 600 adult patients with urothelial bladder cancer. Patients who were diagnosed with urothelial bladder cancer and satisfy the additional eligibility criteria as assessed by the investigator will be invited to participate during routine clinical visit. Only patients who will give their written informed consent will be included. Consecutive patients included in the study will form three study cohorts of equal size (around 200 participants each) according to the stages of urothelial bladder cancer at the time of study inclusion: high-risk NMIBC, MIBC, and mBC.

The investigator will enter medical data of the enrolled patients into the electronic case report form (eCRF) from the source medical documentation. No follow-up is planned, the study will consist of only one visit carried out according to routine clinical practice, where patient's demographic and clinical characteristics as well as medical history and used treatment approaches will be recorded, and formalin-fixed paraffin-embedded (FFPE) tumour tissue samples collected as part of routine clinical practice will be shipped to the central laboratory.

The overall expected duration of the study enrollment is about 18 months or until 600 patients will be included in the study, and all required data (including results of IHC testing in central laboratory) will be collected, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Signed ICF, including consent for FFPE tumor tissue sample testing;
* Confirmed diagnosis of urothelial bladder cancer at NMIBC, MIBC, or mBC stage at study entry;
* For patients with NMIBC: 1. TURBT performed at least 1 month but not more than 12 months prior to study entry; 2. Presence of ≥1 high-risk feature:

  * T1 tumor
  * High grade/G3 tumor
  * CIS (carcinoma in situ)
  * Multiple and recurrent and large (with diameter of largest tumor ≥3 cm) tumors (all conditions must be met in this point);
* For patients with MIBC: Сystectomy performed at least 2 months but not more than 12 months prior to study entry;
* For patients with mBC: mBC diagnosed during 12 months prior to study entry;
* Availability of medical history data;
* Availability of FFPE tumour tissue sample obtained during biopsy and/or surgery.

Exclusion Criteria:

• Participation in any interventional trial since the urothelial bladder cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned study population consists of approximately 600 adult patients with urothelial bladder cancer. Patients who were diagnosed with urothelial bladder cancer and satisfy the additional eligibility criteria as assessed by the investigator will be invited to participate during routine clinical visit. Only patients who will give their written informed consent will be included. Consecutive patients included in the study will form three study cohorts of equal size (around 200 participants each) according to the stages of urothelial bladder cancer at the time of study inclusion: high-risk NMIBC, MIBC, and mBC.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving any intravesical treatment among patients with high-risk NMIBC | 24 months
  Proportion of patients receiving any intravesical treatment among patients with high-risk Non-muscle invasive bladder cancer (ongoing and anamnestic);
Proportion of patients receiving intravesical chemotherapy among patients with high-risk NMIBC | 24 months
  Proportion of patients receiving intravesical chemotherapy among patients with high-risk ongoing and anamnestic Non-muscle invasive bladder cancer (overall and by each treatment regimen);
Proportion of patients receiving intravesical BCG treatment among patients with high-risk NMIBC | 24 months
  Proportion of patients receiving intravesical Bacillus Calmette-Guérin treatment among patients with high-risk ongoing and anamnestic Non-muscle-invasive bladder cancer (overall and by each treatment regimen: induction/ induction + maintenance);
Proportion of patients receiving any intravesical treatment among patients with non-high-risk NMIBC | 24 months
  Proportion of patients receiving any intravesical treatment among patients with non-high-risk Non-muscle-invasive bladder cancer (anamnestic);
Proportion of patients receiving intravesical chemotherapy among patients with non-high-risk anamnestic NMIBC | 24 months
  Proportion of patients receiving intravesical chemotherapy among patients with non-high-risk anamnestic Non-muscle-invasive bladder cancer (overall and by each treatment regimen);
Proportion of patients receiving intravesical BCG treatment among patients with non high-risk anamnestic NMIBC | 24 months
  Proportion of patients receiving intravesical Bacillus Calmette-Guérin treatment among patients with non high-risk anamnestic Non-muscle-invasive bladder cancer(overall and by each treatment regimen: induction/ induction + maintenance);
Proportion of patients without intravesical NMIBC treatment | 24 months
  Proportion of patients without intravesical Non-muscle-invasive bladder cancer (ongoing and anamnestic) treatment (high-risk, non-high-risk)
Number of relapses in high risk NMIBC patients (ongoing and anamnestic) overall and by each treatment regimen | 24 months
  Number of relapses in high risk Non-muscle-invasive bladder cancer patients (ongoing and anamnestic) overall and by each treatment regimen (intravesical chemotherapy, intravesical BCG (induction or induction with maintenance))
Number of relapses in non-high risk NMIBC patients overall and by each treatment regimen, intravesical BCG | 24 months
  Number of relapses in non-high risk Non-muscle-invasive bladder cancer patients (anamnestic) overall and by each treatment regimen (intravesical chemotherapy, intravesical Bacillus Calmette-Guérin (induction or induction with maintenance))
Time to first relapse of NMIBC | 24 months
  Time to first relapse of NMIBC (ongoing and anamnestic)
Proportion of patients receiving neoadjuvant treatment among patients with MIBC | 24 months
  Proportion of patients receiving neoadjuvant treatment among patients with Muscle-invasive bladder cancer (ongoing and anamnestic) (overall and by each treatment regimen);
Rate of pathologic complete response among MIBC patients receiving neoadjuvant treatment | 24 months
  Rate of pathologic complete response among Muscle-invasive bladder cancer patients (ongoing and anamnestic) receiving neoadjuvant treatment (overall and by each treatment regimen);
Proportion of MIBC patients not received neoadjuvant treatment before radical cystectomy | 24 months
  Proportion of Muscle-invasive bladder cancer patients (ongoing and anamnestic) not received neoadjuvant treatment before radical cystectomy.
Proportion of patients received adjuvant treatment among patients with MIBC | 24 months
  Proportion of patients received adjuvant treatment among patients with Muscle-invasive bladder cancer (ongoing and anamnestic) (overall and by each treatment regimen);
Proportion of MIBC patients (anamnestic) received trimodal therapy | 24 months
  Proportion of Muscle-invasive bladder cancer patients (anamnestic) received trimodal therapy (maximal Transurethral resection of bladder tumor + chemoradiation therapy);
Time to progression to mBC from NMIBC and MIBC | 24 months
  Time to progression to metastatic bladder cancer (anamnestic) from Non-muscle-invasive bladder cancer and Muscle-invasive bladder cancer;
Type of progression to mBC from NMIBC and MIBC | 24 months
  Type of progression to Metastatic bladder cancer (anamnestic) from Non-muscle-invasive bladder cancer and Muscle-invasive bladder cancer(localization of metastases);
Proportion of patients with locoregional progression after cystectomy | 24 months
  Proportion of patients with locoregional progression after cystectomy (Muscle-invasive bladder cancer, anamnestic);
Proportions of patients receiving systemic treatment regimens within first-line therapy among patients with mBC | 24 months
  Proportions of patients receiving systemic treatment regimens within first-line therapy among patients with Metastatic bladder cancer (by each treatment regimen);
Proportion of patients with progression on first line mBC treatment | 24 months
  Proportion of patients with progression on first line Metastatic bladder cancer treatment overall and by each treatment regimen.

SECONDARY OUTCOMES:
Prevalence of IHC-defined HER2-positive status among patients with high-risk NMIBC | 24 months
  Prevalence of immunohistochemically-defined HER2-positive status (defined as proportion of patients with 3+ HER2 protein expression based on immunohistochemistry testing of formalin-fixed paraffin-embedded tumor tissue samples) among patients with high-risk Non-muscle-invasive bladder cancer;
Prevalence of IHC-defined HER2-positive status among patients with MIBC | 24 months
  Prevalence of mmunohistochemically-defined HER2-positive status (defined as proportion of patients with 3+ HER2 protein expression based on immunohistochemistry testing of formalin-fixed paraffin-embedded tumour tissue samples) among patients with Muscle-invasive bladder cancer;
Prevalence of IHC-defined HER2-positive status among patients with mBC; | 24 months
  Prevalence of mmunohistochemically-defined HER2-positive status (defined as proportion of patients with 3+ HER2 protein expression based on immunohistochemistry testing of formalin-fixed paraffin-embedded tumour tissue samples) among patients with mBC;
Concordance of immunohistochemically-defined HER2-positive status among 3 patient cohorts | 24 months
  Concordance of immunohistochemically-defined HER2-positive status (defined as proportion of patients with 3+ HER2 protein expression based on immunohistochemistry testing of formalin-fixed paraffin-embedded tumour tissue samples) among patients with Non-muscle-invasive bladder cancer, muscle-invasive bladder cancer and metastatic bladder cancer in primary tumor samples and metastasis if both available;
Prevalence of PD-L1 positive status among patients with mBC | 24 months
  Prevalence of PD-L1 positive status (defined as proportion of patients with at least one of the following criteria based on IHC testing of Formalin-fixed paraffin-embedded tumour tissue sample: (1) ≥25% PD L1 positive tumor cells; (2) ≥25% PD-L1-positive immune cells if >1% of the tumor area contained such cellular elements; or (3) 100% PD-L1-positive immune cells if 1% of the tumor area contained immune cells) among patients with metastatic bladder cancer.

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (13):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/